CLINICAL TRIAL: NCT01719094
Title: RITHM - Resonance Imaging Trial for Heart Biomarkers in Adolescent/Young (AYA) Cancer Survivors
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00014375; CCCWFU 99312 (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2012-10-30; First posted 2012-11-01 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: if Aortic Stiffness; Myocardial Wall Strain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Childhood Cancer Surviviors
- Adolescent/young adults with no cancer history
- Newly diagnosed cancer patients

SUMMARY:
Cardiovascular events are the leading non-cancer cause of mortality after childhood cancer, occurring at a significantly younger age than in the general population. The increased incidence of cardiovascular events adversely impacts the functional capacity, morbidity, and mortality of otherwise relatively healthy 20 to 40 year old individuals. Moreover, understanding of the mechanisms by which cancer treatment could influence the occurrence of latent cardiovascular events is unavailable. Our group and others have established independent, noninvasive magnetic resonance imaging (MRI) measures of cardiovascular risk in middle aged and elderly individuals. Cardiovascular risk include, acute coronary syndromes, cardiac death, and congestive heart failure. The goal of this application is to show that childhood cancer survivors at risk for impaired cardiovascular and cerebrovascular health have increased aortic stiffness, when compared to healthy adolescent and young adult age mate. Studies are designed to determine if MRI measures of cardiovascular function differ between adolescent/adult childhood cancer survivors (n=60), age matched controls (n=30), and adolescents/young adults with planned treatment with chemo- and radiation therapy (n=25). The investigators propose that MRI markers responsible for cardiovascular events represent new clinical indicators that could be targeted to treat asymptomatic cardiovascular diseases.

ELIGIBILITY:
Inclusion Criteria:

Childhood Cancer Survivors

* Diagnosis of cancer at age 21 or younger
* Current age 16-40 years
* 1year and ≤ 15 years from end of cancer treatment
* Received anthracycline chemotherapy
* Asymptomatic (Appendix VII: absence of palpitations, dyspnea, edema or anginal symptoms)
* No pre-existing diagnosis with regard to cardiovascular or cerebrovascular disease status.

Adolescent/young adults with no cancer history

* No prior diagnosis of cancer, diabetes, or lung disease
* Current age 16-40 years
* No history of radiation to chest or neck
* No prior history of chemotherapy
* Asymptomatic (Appendix VII : absence of palpitations, dyspnea, edema or anginal symptoms) and without a pre-existing diagnosis with regard to cardiovascular or cerebrovascular disease status.

Newly diagnosed cancer patients

* Diagnosis of cancer at age 25 or younger
* Current age 7-25 years
* Planned receipt of anthracycline chemotherapy
* Planned treatment course ≤ 15 months
* No pre-existing cardiovascular disease

Exclusion Criteria:

All groups

* Subjects with implanted electronic devices, including but not limited to: pacemakers, defibrillators, functioning neurostimulator devices, or other implanted electronic devices
* Subjects with ferromagnetic cerebral aneurysm clips, or other intraorbital/intracranial metal
* Claustrophobia
* Subjects who received total body irradiation or cranial irradiation
* History of acute myocardial infarction
* Significant ventricular arrhythmias (>20 PVC's/minute due to gating difficulty)
* Medical history of moderate or severe aortic stenosis, or other significant valvular disease
* Women who are pregnant
* Those with pre-existing history (by self report in Group B and review of medical records in addition to self-report for Groups A & C) of abnormal cardiovascular function including: congenital heart disease, hypertension, diabetes, hypercholesterolemia on treatment, a body mass index >35, history of asymptomatic cardiac dysfunction (defined as an ejection fraction < 40 and/or shortening fraction < 28) or symptomatic cardiac dysfunction (congestive heart failure), stroke, renal dysfunction by history/medical records (serum creatinine >1.4), anemia, obstructive or restrictive airways disease
* Asymptomatic cardiac dysfunction (defined as an ejection fraction < 40 and/or shortening fraction < 28 on last ECHO or MUGA)
* Participants unwilling to complete the protocol (1 visit for Group A, B; 3 scan studies for Group C)
* Participants unable to provide informed consent via a guardian or self

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Childhood cancer survivors, adolescent/young adults with no cancer history and newly diagnosed cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2012-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
To determine if aortic stiffness or myocardial wall strain is increased in childhood cancer survivors who received anthracycline chemotherapy | Day 1

SECONDARY OUTCOMES:
To determine if aortic stiffness changes during treatment with anthracycline chemotherapy in childhood cancer patients | approximately 6 months
  n=25

CONTACTS AND LOCATIONS:
Overall Officials: Sharon M Castellino, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - Emory University School of Medicine, Atlanta, Georgia
  - Wake Forset University Health Sciences, Winston-Salem, North Carolina